CLINICAL TRIAL: NCT04279249
Title: Home Air Filtration for Traffic-Related Air Pollution
Acronym: HAFTRAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Somerville Transportation Equity Partnership, Inc. (Unknown); Tufts University (Other); Olin College of Engineering (Unknown); Welcome Project Inc (Unknown); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Douglas Brugge, Professor, UConn Health
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 20-109-2; 1R01ES030289 (NIH)
Record Dates: First submitted 2019-09-10; First posted 2020-02-21 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2023-06

CONDITIONS: Cardiovascular Risk Factor; Blood Pressure
Keywords: Ultrafine Particles (UFP); HEPA; Traffic-Related Air Pollution; Air Filtration; In-home

STUDY DESIGN:
Intervention Model Description: This study is a randomized crossover trial, in which study participants are randomly assigned (by computer) to different arms of the study in which they receive different interventions - in this case, either the HEPA air filter or the sham filter. The two arms will run concurrently, rather than sequentially.
  Primary Outcome Measures will be measured concurrently, rather than at separate time points (i.e., blood pressure and blood samples will both be taken at study onset, 30 days, 60 days and 90 days) and therefore fall within the same time points.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HEPA Filtration (Active Comparator)
  Interventions: Other: HEPA Air Filtration
- Sham HEPA Filtration (Sham Comparator)
  Interventions: Other: Sham HEPA Air Filtration

INTERVENTIONS:
Other: HEPA Air Filtration — 2 HEPA air filters placed in home (one in bedroom, one in living room) for 30 days
  Arms: HEPA Filtration
Other: Sham HEPA Air Filtration — 2 HEPA air filter devices with filter removed placed in home (one in bedroom, one in living room) for 30 days
  Arms: Sham HEPA Filtration

SUMMARY:
This study is a blinded randomized crossover efficacy trial (N=172 households consisting of 207 participants) of High Efficiency Particulate Air (HEPA) filtration in near-highway homes that lack mechanical air-handling systems. Households will be randomized to 30 days of either filtration or sham filtration followed by a 30 washout period with a subsequent 30-day period of the alternative assignment. Room air filters that are commercially available will be placed in the bedroom and living room of each home.

The investigators will measure UFP and PM2.5 concentrations in 20% of the homes during filtration and sham periods and assess personal exposure in a subset of participants. The investigators will also assess chemical composition of particulate air pollution in 10 homes/year for exploratory purposes that could lead to future lines of research. The primary health endpoints will be participants' hsCRP and peripheral blood pressure, measures that the investigators have used in multiple observational studies of UFP as well as in pilot filtration intervention studies. Secondary biological measures that contribute to understanding biological pathways will be IL-6 (inflammation), D-dimer (coagulation), metabolome, central pressure and arterial stiffness. The primary intention to treat analysis will compare outcomes between HEPA filtration to sham filtration. The investigators will have 80% power to detect a difference of 0.6 mg/L in change in hsCRP and a difference in reduction in systolic blood pressure of 3.5 mmHg compared to participants who receive no filtration. Having participants serve as their own controls in the within-subject comparisons of intervention effectiveness increases statistical power and eliminates the possibility of baseline imbalances in demographic and clinical characteristics. A social science evaluation will inform final adjustments to the investigators' approach at the start and also assess participant acceptance and experience with the intervention at the end. The investigators' primary innovation is that this will be the first near highway HEPA intervention trial that is large enough and careful enough to be policy-relevant.

DETAILED DESCRIPTION:
Specific Aims:

Specific Aim 1: To test the effect of HEPA filtration on markers of cardiovascular risk for adults who live near urban highways. 207 participants will be enrolled in a double blind, randomized crossover trial of 30-day periods with and without filtration separated by a 30-day wash out period. The intervention will be during colder months (Oct-Mar) when ambient UFP are elevated and windows tend to be closed, thereby allowing for maximization of the exposure contrast between HEPA and sham conditions. The investigators hypothesize that the HEPA filtration intervention will be associated with indications of improved health in the primary health outcomes: blood pressure (systolic, diastolic, and pulse pressure); and hsCRP (a measure of inflammation).

Specific Aim 2: To assess whether the intervention succeeded or failed in participant homes. To determine effectiveness of the filtration intervention, the investigators will 1) measure particle pollution levels inside and outside 20% of the homes, and 2) use quantitative surveys and open-ended questions to evaluate how participants interacted with the intervention.

Specific Aim 3: To assess biomarkers that can suggest biological pathways by which filtration affects cardiovascular risk. Study participants will be measured for IL-6 (inflammation), D-dimer (coagulation), central blood pressure, and arterial stiffness (endothelial dysfunction), which constitute key steps along the presumed biological pathways. The peripheral blood plasma of all participants will also undergo metabolome analysis to provide additional evidence of biological pathways. The investigators propose this to follow on an exciting recent study that used a similar approach 24, and preliminary metabolome analysis.

Exploratory Aims: To analyze particle composition. In a subset of homes (30 homes total, 10/year), the investigators will perform detailed physical and chemical analysis of PM1 (particles <1,000 nm) to inform future work on composition-dependent health impacts and filtration effectiveness for UFP. Also in a subset of homes, assess personal exposures for 24 participants. The scientific premise is that HEPA filtration in homes without mechanical ventilation systems can reduce UFP (and overall PM) levels leading to positive changes in biomarkers. The study design and approach are rigorous, using a double blind, randomized cross over trial. The investigators will also measure objective biomarkers of risk of cardiovascular disease. The primary innovation is that this will be the first HEPA intervention trial near highways that is large enough to rule in or out efficacy of stand-alone HEPA filters from traffic pollution

Hypotheses:

1. For Aim 1, the investigators hypothesize that the HEPA filtration intervention will be associated with statistically significant improvements of peripheral blood pressure (BP) and C-reactive protein (hsCRP).
2. The investigators hypothesize that measures collected for Aim 3 will show that UFP is associated with antioxidant pathways, in vivo generation of reactive oxygen species, and processes critical to endothelial functions, as well as indicators of early vascular aging.

ELIGIBILITY:
Inclusion Criteria:

* residence within 200 m of interstate I-93 in Somerville
* live at home full time
* cognitive ability to answer questionnaires
* able to speak English/Spanish

Exclusion Criteria:

* in-home mechanical air handling system with forced air pushed through vents
* smoker or lives with smoker(s)
* history of heart attack, stroke, or other major cardiovascular outcome
* taking anti-hypertensive or anti-inflammation medications
* occupational or other routine high exposures (away from home) to traffic pollution
* extensive use of candles/incense inside the home

Preferred Criteria:

* residents of apartments with highway-facing windows and that are no more than 3 stories tall

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure at 1 Month | measured at study onset and 30 days
  Seated blood pressure measured using ambulatory monitors
Change in High Sensitivity C-Reactive Protein (hsCRP) at 1 Month | blood sample taken at study onset and 30 days
  inflammation marker assayed from blood samples

SECONDARY OUTCOMES:
Change in D-dimer at 1 Month | blood sample taken at study onset and 30 days
  coagulation marker assayed from blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Doug Brugge, PhD, Principal Investigator — Tufts University
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh-Smith K, Sprague Martinez L, Eliasziw M, Lerman Ginzburg S, Hudda N, Betz GM, Gurcan A, Vazquez-Dodero T, Mertl A, Goldstein-Gelb W, Zamore W, Brugge D. Reaction to at-home air purifiers installed to reduce traffic-related air pollution in near-highway residences. Trials. 2024 Aug 19;25(1):551. doi: 10.1186/s13063-024-08388-z. PMID 39160612